CLINICAL TRIAL: NCT04074525
Title: Delivery Decisions in Extreme Prematurity: Evaluating Decisional Regret
Brief Title: Evaluating Decisional Regret Among Mothers
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Collaborators: Providence Health & Services (Other)
Responsible Party: Sponsor
Other Study IDs: DDD604440
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Extreme Prematurity; Birth, Preterm; Pregnancy Preterm
Keywords: Decisional regret; Comfort care; Palliative care; Infant resuscitation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The anticipated birth of an extremely low gestational age infant presents many complex and ethically challenging questions, including whether to initiate resuscitation or comfort care after delivery. Failure to identify and align decision-making to parents' values during periviabilty counseling may result in greater opportunity for decisional regret. The goal of the proposed research is to assess decisional regret in mothers of extremely premature births and to compare decisional regret in mothers who chose resuscitation at time of delivery to those who chose comfort care. Approximately 1000 mothers of infants born extremely premature at 2 perinatal centers in the US will be surveyed.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of infants born between 22 and 25 completed weeks gestation during the study timeframe.
* Mothers who had a documented perinatal consult
* Greater than 18 years old

Exclusion Criteria:

* Potential life limiting fetal diagnoses aside from prematurity and non-English primary language

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender eligibility for this study will be determined by women who had the ability to become pregnant and give birth at one of 2 perinatal centers.
Study Population: The study population will consist of mothers who delivered infants between 22 and 25 completed weeks gestation during the study timeframe at one of two US perinatal centers.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Decisional regret | Within the last 14 years
  To assess decisional regret in mothers of extremely premature liveborn infants.
Comparison of decisional regret | Within the last 14 years
  Comparison of decisional regret in mothers who chose resuscitation versus mothers who chose comfort care at the time of delivery.

SECONDARY OUTCOMES:
Define characteristics associated with decisional regret | Within the last 14 years
  Identify characteristics, and specifically potentially modifiable characteristics, that are associated with decisional regret in our population of mothers.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Belden, DO, Principal Investigator — Christiana Care Health Services, Inc.
Locations (1):
- Christiana Care Health Services, Inc., Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belden L, Kaempf J, Mackley A, Kernan-Schloss F, Chen C, Sturtz W, Tomlinson MW, Guillen U. Evaluating decision regret after extremely preterm birth. Arch Dis Child Fetal Neonatal Ed. 2025 Feb 21;110(2):191-199. doi: 10.1136/archdischild-2024-327287. PMID 39164062